CLINICAL TRIAL: NCT03242551
Title: The Role of Multimodal Imaging and Circulating Biomarkers in Predicting the Response of Neoadjuvant Chemotherapy for Breast Cancer
Brief Title: Biomarkers Investigation of Neoadjuvant Chemotherapy for Breast Cancer
Acronym: BINC-B
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Principal Investigator, Wenyong Tan, Director, Shenzhen People's Hospital
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Shenzhen BC-001
Record Dates: First submitted 2017-07-28; First posted 2017-08-08 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: epirubicin, paclitaxol, cyclophosphamide, trastuzumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant chemotherapy (Experimental): Epirubicin 100mg/m2 and cyclophosphamine 600mg/m2 for four cycles followed by paclitaxol 175mg/m2 for four cycles with (for patients with positive HER-2) or without Trastuzumab (loading dose of 6 mg/kg followed by 4 mg/kg every 2 weeks for four cycles), each cycle is 14 days.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — "AC" followed by "T" Chemotherapy with or without trastuzumab, i.e. Epirubicin 100mg/m2 and cyclophosphamine 600mg/m2 for four cycles followed by paclitaxol 175mg/m2 for four cycles with (for patients with positive HER-2) or without Trastuzumab (loading dose of 6 mg/kg followed by 4 mg/kg every 2 weeks for four cycles), each cycle is 14 days.

SUMMARY:
The BINC-B trial is a diagnostic and interventional study in which various function imaging methods as Magnetic Resonance Imaging (PWI, DWI and DCE-MRI) and will be compared with common imaging methods (mammography and/or ultrasound) to investigate if an early response to a combined neoadjuvant chemotherapy in operable or potentially operable breast cancer. For breast cancer patients with positive HER-2, additional Herceptin could improve the response further. In this study the efficacy of combined neoadjuvant therapy with or without Herceptin should be evaluated and the role in predicting the tumor response with different imaging should be estimated.

DETAILED DESCRIPTION:
Firstly, the investigators aim to show that the results of functional imaging including dynamic enhanced, diffuse weighted, and perfusion MR imaging biomarkers as well the ultrasonic outcome could be used to predict the response to the neoadjuvant chemotherapy for operable and potentially operable breast cancer (luminal B, HER-2 positive and triple negative).

Secondly, the investigators will study the role of peripheral blood biomarker including circulating tumor DNA (ctDNA), circulating endothelial cells (CECs) and subsets, myeloid-derived suppressor cells (MDSCs), and lymph cell subsets and their combinations could predict the response of the tumor measured with imaging.

Thirdly, the investigators will establish a mode with these multiple imaging and serum biomarker panel as well as their changes during the treatment course establish to predict the response to neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria

* Age ≥18 years and ≤70 years
* Female
* Operable or potentially operable primary breast cancer (≥ cT2, N0 or N+, M0);
* Confirmed by core biopsy
* Histological confirmed unilateral, solitaire breast cancer
* Baseline LVEF ≥55% (measured by echocardiography) according to institution specific norm
* Informed consent for clinical trial including analysis of predictive imaging tests and biomarkers
* Clinically or by imaging (mammogram, MRI or US) assessed breast cancer ≥2 cm with bi-dimensional measurable lesion independent of nodal status
* Negative pregnancy test (urine or serum) within 7 days prior to registration if patient is premenopausal with intact reproductive organs and if patient is less than one year after menopause
* ECOG Performance status 0-2
* Adequate organ function for cytotoxic chemotherapy
* Adequate renal function including Serum creatinine ≤ ULN, Measured or calculated creatinine clearance > 60 ml per min
* Absolute neutrophil count ≤ 1500/µL, platelet count ≥ 100,000/µL
* Bilirubin ≤ ULN; ALT or AST ≤ 1.5 x ULN, and alkaline phosphatase ≤2.5 x ULN
* Patients must be available and compliant for treatment and follow-up

Exclusion Criteria

* Evidence of distant metastases by clinical or imaging diagnosis
* Multifocal primary tumor, defined as histologically confirmed tumor-manifestations within different quadrants; distance ≥ 4 cm
* Pre-existing motor or sensory neuropathy of a severity ≥ grade 2 NCI criteria
* Previous breast cancer
* Prior malignancy with a disease-free survival of < 5 year
* Prior malignancy which has not been curatively treated
* Inflammatory breast cancer
* Prior systemic therapy for cancer
* Patients with immunosuppressive therapy
* Pregnant or lactating women
* Women of childbearing potential not using highly effective birth control
* Patients with known hypersensitivity reactions to the compounds or incorporated substances of trastuzumab or its constituents (for HER2+ tumors)
* Invasive malignancy which could affect compliance with the protocol or interpretation of results
* Other serious illness or medical condition including: Known or suspected congestive heart failure (>NYHA I) and/or coronary heart disease, Angina pectoris requiring antianginal medication; Previous history of myocardial infarction, Evidence of transmural infarction on ECG, Un- or poorly controlled arterial hypertension (i.e. BP >150/100 mmHg under treatment with two antihypertensive drugs), Rhythm abnormalities requiring permanent treatment; Clinically significant valvular heart disease, Patients with dyspnea at rest due to malignant or other disease or who require supportive oxygen therapy, Active serious uncontrolled infections, Poorly controlled diabetes, History of hypertensive crisis or hypertensive encephalopathy; History of TIA or CVA
* Neutrophil count of < 1500, platelet count of < 100,000/µL, Haemoglobin < 10 g/dL
* Inadequate bone marrow, hepatic and renal functions as evidenced by the following: Serum total bilirubin > ULN, ALT or AST > 1.5 x ULN, Alkaline phosphatase > 2.5 x ULN, serum creatinine > ULN
* Concurrent treatment with any other anti-cancer therapy
* No informed consent for analysis of predictive imaging tests and biomarkers
* Contraindications against MRI: Cardiac pacemakers, other forms of medical or biostimulation implants, ferromagnetic foreign bodies or metallic implants (e.g. surgical protheses, aneurysm clips), implanted insulin pumps, valvular implants, allergy to contrast agent, renal insufficiency, claustrophobia
* Active peptic ulcer, incomplete wound healing or unhealed bone fracture
* Disease significantly affecting gastrointestinal function, e.g. malabsorption syndrome, resection of the stomach or small bowel, ulcerative colitis, abdominal fistula, intra-abdominal abscess within 6 months of enrolment or gastrointestinal perforation
* Concurrent treatment with other experimental drugs; participation in another clinical trial with any investigational drug within 30 days prior to study entry
* Chronic daily treatment with corticosteroids (dose of > 10 mg/day methylprednisolone equivalent) (excluding inhaled steroids)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-11-08 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) | from the first day of the the first cycle (each cycle is 14 days) of neoadjuvant chemotherapy to the date that breast and axillary sugery will be performed
  Rate of pathological complete response (pCR) following neoadjuvant therapy and to determine efficacy of neoadjuvant therapy in primary breast cancer using pCR (According to National Surgical Adjuvant Breast and Bowel Project guideline)

SECONDARY OUTCOMES:
Response rate | from the first day of the the first cycle (each cycle is 14 days) of neoadjuvant chemotherapy to the date that breast and axillary sugery will be performed
  the summary of clinical complete response and partial response (RESICIST 1.1 criteria)
Disease free survival | from the first day of the the first cycle of neoadjuvant chemotherapy (each cycle is 14 days) to the date of first documented progression or date of death from breast cancer, whichever came first, assessed up to 60 months
  from the beginning of neoadjuvant chemotherapy to the confirmed time of recurrence or metastatic disease, or death due to any other cause.
Overall survival | from the first day of the the first cycle (each cycle is 14 days) of neoadjuvant chemotherapy to the date of death from any cause, whichever came first, assessed up to 60 months
  from the beginning of neoadjuvant chemotherapy to the death with any causes

CONTACTS AND LOCATIONS:
Overall Officials: Wenyong Tan, Dr., Principal Investigator — Shenzhen People Hospital
Locations (2):
- China (2):
  - Department of Oncology, Shenzhen, Guangdong
  - Shenzhen People Hospital, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: Yes
all the individual data will be open to the other researchers
Supporting Information: Study Protocol, CSR
Time Frame: After the data is formally published
Access Criteria: open acess

REFERENCES:
- [Background] Marinovich ML, Sardanelli F, Ciatto S, Mamounas E, Brennan M, Macaskill P, Irwig L, von Minckwitz G, Houssami N. Early prediction of pathologic response to neoadjuvant therapy in breast cancer: systematic review of the accuracy of MRI. Breast. 2012 Oct;21(5):669-77. doi: 10.1016/j.breast.2012.07.006. Epub 2012 Aug 3. PMID 22863284
- [Background] Prevos R, Smidt ML, Tjan-Heijnen VC, van Goethem M, Beets-Tan RG, Wildberger JE, Lobbes MB. Pre-treatment differences and early response monitoring of neoadjuvant chemotherapy in breast cancer patients using magnetic resonance imaging: a systematic review. Eur Radiol. 2012 Dec;22(12):2607-16. doi: 10.1007/s00330-012-2653-5. Epub 2012 Sep 16. PMID 22983282
- [Background] Braman NM, Etesami M, Prasanna P, Dubchuk C, Gilmore H, Tiwari P, Plecha D, Madabhushi A. Erratum to: Intratumoral and peritumoral radiomics for the pretreatment prediction of pathological complete response to neoadjuvant chemotherapy based on breast DCE-MRI. Breast Cancer Res. 2017 Jul 10;19(1):80. doi: 10.1186/s13058-017-0862-1. No abstract available. PMID 28693537
- [Background] Murtaza M, Dawson SJ, Tsui DW, Gale D, Forshew T, Piskorz AM, Parkinson C, Chin SF, Kingsbury Z, Wong AS, Marass F, Humphray S, Hadfield J, Bentley D, Chin TM, Brenton JD, Caldas C, Rosenfeld N. Non-invasive analysis of acquired resistance to cancer therapy by sequencing of plasma DNA. Nature. 2013 May 2;497(7447):108-12. doi: 10.1038/nature12065. Epub 2013 Apr 7. PMID 23563269
- [Background] Morganella S, Alexandrov LB, Glodzik D, Zou X, Davies H, Staaf J, Sieuwerts AM, Brinkman AB, Martin S, Ramakrishna M, Butler A, Kim HY, Borg A, Sotiriou C, Futreal PA, Campbell PJ, Span PN, Van Laere S, Lakhani SR, Eyfjord JE, Thompson AM, Stunnenberg HG, van de Vijver MJ, Martens JW, Borresen-Dale AL, Richardson AL, Kong G, Thomas G, Sale J, Rada C, Stratton MR, Birney E, Nik-Zainal S. The topography of mutational processes in breast cancer genomes. Nat Commun. 2016 May 2;7:11383. doi: 10.1038/ncomms11383. PMID 27136393